CLINICAL TRIAL: NCT05651035
Title: Effects of Breastfeeding and Bottle Feeding as the Initial Oral Feeding on Physiological Parameters and Feeding Performance in Preterm Infants: A Randomized Controlled Study
Brief Title: Breastfeeding and Bottle Feeding: Impact on Preterm Infants' Physiology and Feeding Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nagihan Sabaz, Principal Investigator, Research Assistant, PhD candidate, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10840098-604.01.01-E.14287
Record Dates: First submitted 2022-11-29; First posted 2022-12-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Preterm; Breastfeeding; Bottlefeeding; Premature
Keywords: preterm infants; oral feeding; breastfeeding; bottlefeeding; physiological parameters; test weighing; initial oral feeding; Neonatal Intensive Care Unit; Cue-Based oral feeding; Transition to oral feeding
MeSH Terms: conditions — Premature Birth; Breast Feeding; Bottle Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breastfeeding group (Experimental): Preterm infants in this group are breastfed by their mothers during their first oral feeding. Before, during and after feeding, the preterm infant's oxygen saturation level and peak heart rate are measured for 30 minutes. In addition, the test test weighing is determined by weighing the baby before and after feeding.
  Interventions: Other: oral feeding
- Bottle-feeding group (No Intervention): Preterm infants in this group are fed with their mother's milk in the bottle during their first oral feeding.

INTERVENTIONS:
Other: oral feeding — In experimental group infants: Preterms in this group will be breastfed by their own mother.
  In control group infants: Preterms in this group will be fed by the researcher by putting the baby's own mother's milk in the bottle. During feeding, the preterm will be placed on the lap by the researcher in a standing position on the same mother's breast, and will be given a raised side-lying position. In this position, the preterm's head and body will be elevated 45-60 degrees with the help of a small pillow. While the researcher will support the preterm's head, neck and shoulder with one hand, he will control the bottle with the other hand. By touching the preterm's nipple to the preterm's lips, the preterm will be prepared for feeding, and the bottle will be placed in the baby's mouth with the mouth opening and the tongue lowering. During feeding, stimulating movements such as pushing the bottle back and forth in the mouth, which will lead the newborn to suck faster, will not be made.
  Arms: Breastfeeding group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of breastfeeding on the infant's test weight and physiological characteristics (oxygen saturation and heart rate) in preterm infants in the Neonatal Intensive Care Unit during the transition to oral feeding.

The main question it aims to answer are:

• Is there a difference in test weight and physiological parameters between the infants in whom the first oral feeding was performed by the mother and the infants in whom the first oral feeding was performed by the intensive care unit nurse with a bottle? Researchers will compare the breastfed group with the bottle-fed group to see if there are differences in test weight and physiological parameters.

DETAILED DESCRIPTION:
In the pre-feeding stage of the research, the parents of the preterms included in the sample will be met and informed about the research. Written and verbal consent will be obtained from parents who agreed to participate in the study. "Preterm Infants Information Form" will be filled by the researcher before feeding and "Feeding Monitoring Form" will be filled during feeding. By randomization, it will be determined which of the experimental and control groups the preterm infant will be assigned to. It will be ensured that the interventions that will affect the vital signs of the preterms in both groups before feeding are not applied. Oxygen saturation and heart rate will be monitored for 30 minutes before, during and after feeding for all groups. Preterms in both groups will be dressed in clean and dry diapers by cleaning their bottoms before feeding, and will be weighed naked with a digital baby scale by removing their clothes. Weighing the preterms with an electronic precision balance before and after feeding - the test weighing - will be used to measure the amount of milk the preterm is expressing from the breast or bottle. The preterm will then be fed loosely wrapped in a cotton blanket. If the oxygen saturation level of all preterm infants falls below 90% during feeding, it will be considered desaturated and the feeding will be stopped. The preterm infants will continue to be fed when the oxygen saturation is ≥ 90% and the heart rate is 120-160/min. Feeding will be limited to a total of 30 minutes for infants in both groups, including rest intervals, and will not take longer. When the feeding is complete, preterms in both groups will be weighed naked without changing the diaper under the feeding process. It will be ensured that interventions that may affect the vital signs of all preterms included in the study are not applied when feeding is completed. The oxygen saturation and heart rate of the preterms in both groups will be monitored for 30 minutes after the feeding is completed. When feeding is complete, preterms in both groups will be placed on the same mother's breast in the right lateral position to facilitate gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* Gestation week at birth determined according to the mother's last menstrual date is 26-31+6 weeks,
* Postmenstrual week at the time of the study was 32-36+6 weeks,
* Having a body weight of 1500 grams or more at the time of inclusion in the study,
* Suggested by the physician to switch to oral nutrition and switched from enteral nutrition to oral nutrition for the first time,
* Breastfed,
* Preterm infants whose parents' consent was obtained for inclusion in the study and whose parents signed the informed consent form

Exclusion Criteria:

* Receiving oxygen,
* Craniofacial anomalies such as cleft palate, cleft lip, facial muscle paralysis,
* Preterm infants with any gastrointestinal, neurological and genetic disease (necrotizing enterocolitis, third and fourth level intracranial hemorrhage, periventricular leukomalacia, hydrocephalus, down syndrome, omphalocele, non-gastrodeia, short bowel syndrome and other diseases)

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
preterm infant's weight gain | 30 minutes before oral feeding and 30 minutes after oral feeding is complete
  It is to determine the weight gain by weighing the preterm infant with the same diaper before and after oral feeding.

SECONDARY OUTCOMES:
Oxygen saturation | 30 minutes
  Oxygen saturation ≥ 90% during and just after oral feeding
Heart rate | 30 minutes
  Heart rate 120-160/min during and just after oral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Gözen, Ph.D., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- IstanbulUC, Avcılar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girgin BA, Gozen D, Karatekin G. Effects of two different feeding positions on physiological characteristics and feeding performance of preterm infants: A randomized controlled trial. J Spec Pediatr Nurs. 2018 Apr;23(2):e12214. doi: 10.1111/jspn.12214. Epub 2018 Mar 5. PMID 29504676
- [Background] Chen CH, Wang TM, Chang HM, Chi CS. The effect of breast- and bottle-feeding on oxygen saturation and body temperature in preterm infants. J Hum Lact. 2000 Feb;16(1):21-7. doi: 10.1177/089033440001600105. PMID 11138220
- [Background] Fontana C, Menis C, Pesenti N, Passera S, Liotto N, Mosca F, Roggero P, Fumagalli M. Effects of early intervention on feeding behavior in preterm infants: A randomized controlled trial. Early Hum Dev. 2018 Jun;121:15-20. doi: 10.1016/j.earlhumdev.2018.04.016. Epub 2018 May 3. PMID 29730130
- [Background] Goldfield EC, Richardson MJ, Lee KG, Margetts S. Coordination of sucking, swallowing, and breathing and oxygen saturation during early infant breast-feeding and bottle-feeding. Pediatr Res. 2006 Oct;60(4):450-5. doi: 10.1203/01.pdr.0000238378.24238.9d. Epub 2006 Aug 28. PMID 16940236
- [Background] Gianni ML, Sannino P, Bezze E, Comito C, Plevani L, Roggero P, Agosti M, Mosca F. Does parental involvement affect the development of feeding skills in preterm infants? A prospective study. Early Hum Dev. 2016 Dec;103:123-128. doi: 10.1016/j.earlhumdev.2016.08.006. Epub 2016 Aug 31. PMID 27591506
- [Background] Rocha NM, Martinez FE, Jorge SM. Cup or bottle for preterm infants: effects on oxygen saturation, weight gain, and breastfeeding. J Hum Lact. 2002 May;18(2):132-8. doi: 10.1177/089033440201800204. PMID 12033074
- [Background] Moral A, Bolibar I, Seguranyes G, Ustrell JM, Sebastia G, Martinez-Barba C, Rios J. Mechanics of sucking: comparison between bottle feeding and breastfeeding. BMC Pediatr. 2010 Feb 11;10:6. doi: 10.1186/1471-2431-10-6. PMID 20149217
- [Background] Stevens EE, Gazza E, Pickler R. Parental experience learning to feed their preterm infants. Adv Neonatal Care. 2014 Oct;14(5):354-61. doi: 10.1097/ANC.0000000000000105. PMID 25000100
- [Background] Thoyre SM, Pados BF, Shaker CS, Fuller K, Park J. Psychometric Properties of the Early Feeding Skills Assessment Tool. Adv Neonatal Care. 2018 Oct;18(5):E13-E23. doi: 10.1097/ANC.0000000000000537. PMID 30239407
- [Background] Settle M, Francis K. Does the Infant-Driven Feeding Method Positively Impact Preterm Infant Feeding Outcomes? Adv Neonatal Care. 2019 Feb;19(1):51-55. doi: 10.1097/ANC.0000000000000577. PMID 30672812
- [Derived] Sabaz N, Gozen D, Tastekin A. Effects of breastfeeding and bottle feeding as the initial oral feeding on physiological parameters and feeding performance in preterm infants: A randomized controlled study. J Pediatr Gastroenterol Nutr. 2025 Nov 29. doi: 10.1002/jpn3.70295. Online ahead of print. PMID 41318959
- See also: Assessment of Oral Feeding Readiness in Preterm Infants — https://www.turkiyeklinikleri.com/article/tr-preterm-bebeklerde-oral-beslenmeye-hazir-oluslugun-degerlendirilmesi-78966.html
- See also: Evidence-Based Interventions Supporting Oral Feeding in Preterm Infants — https://dergipark.org.tr/en/pub/clinexphealthsci/issue/35066/389077